CLINICAL TRIAL: NCT06439251
Title: Effects of Mulligan Technique With or Without Diclofenac Phonophoresis on Pain, Range of Motion and Functional Disability of Knee Joint in Patients With Patellofemoral Pain Syndrome
Brief Title: Effects of Mulligan Technique With or Without Diclofenac Phonophoresis on Patellofemoral Pain Syndrome.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Zunaira saeed, Principal Investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-546-10-2023
Record Dates: First submitted 2024-02-27; First posted 2024-06-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain Syndrome,; Mulligan mobilization; Phonophoresis; diclofenac
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diclofenac Phonophoresis (Experimental): The participants randomly allocated in Group A were receive the Phonophoresis (Ultrasound with Diclofenac gel for 5 minutes and intensities 1 MHz and 1.5 W/cm² pulsed waves was used in the therapy sessions on affected knee with diclofenac gel on ultrasound head) as experimental technique
  Interventions: Combination Product: Group 1
- Mulligan Technique (Active Comparator): The treatment involved routine physiotherapy with TENS at 80 Hz and a pulse duration of 50-100 μs, followed by a 15-minute hot pack. It also included stretching exercises for the hamstring and calf muscles, isometric strengthening of the quadriceps and VMO, straight leg raises with traction, and tibial gliding techniques. The MWM technique consisted of SLR with traction, repeated 10 times with 3 sets and a 1-minute interval in between.
  Interventions: Combination Product: Group 2

INTERVENTIONS:
Combination Product: Group 1 — The treatment included TENS therapy, hot pack application, stretching exercises, isometric strengthening, straight leg raises with traction, and tibial gliding techniques. Participants in Group A also received Phonophoresis as an experimental technique.
  Arms: Diclofenac Phonophoresis
Combination Product: Group 2 — The treatment included routine physiotherapy with TENS, hot pack application, stretching exercises, isometric strengthening, straight leg raises with traction, and tibial gliding techniques.
  Arms: Mulligan Technique

SUMMARY:
The patellofemoral pain syndrome (PFPS) is a common cause for "anterior knee pain" and mainly affects young women. the effectiveness of Mulligan technique with or without diclofenac phonophoresis on pain, range of motion and functional disability of knee joint in patients with patellofemoral pain syndrome is known little. This study, ethically approved, focused on patients with anterior knee pain referred to the Physical Therapy Department from Lahore General Hospital. After eligibility assessments and consent, participants were randomly assigned to Group A (Experimental) or Group B (Control). Over four weeks, three sessions per week, routine physiotherapy and specific exercises will be administered, with Group A receiving additional Phonophoresis using ultrasound and diclofenac gel. Outcome variables (Numeric Pain Rating Scale, KOOS-PF, Universal Goniometer) will be assessed by a blinded assessor at baseline and study completion.

DETAILED DESCRIPTION:
Background: The patellofemoral pain syndrome (PFPS) is a common cause for "anterior knee pain" and mainly affects young women without any structural changes such as increased Q-angle or significant pathological changes in articular cartilage.

Objective: To evaluate the effectiveness of Mulligan technique with or without diclofenac phonopheresis on pain, range of motion and functional disability of knee joint in patients with patellofemoral pain syndrome.

Methodology: This study, ethically approved, focused on patients with anterior knee pain referred to the Physical Therapy Department from Lahore General Hospital. After eligibility assessments and consent, participants were randomly assigned to Group A (Experimental) or Group B (Control). Over four weeks, three sessions per week, routine physiotherapy and specific exercises were administered, with Group A receiving additional Phonophoresis using ultrasound and diclofenac gel. Outcome variables (Numeric Pain Rating Scale, KOOS-PF, Universal Goniometer) were assessed by a blinded assessor at baseline and study completion.

ELIGIBILITY:
Inclusion Criteria:

* • Patients of age range 20-45 years and both genders (Rehman, 2021 #171)

  * Unilateral anterior knee pain persisting for over two months, referred by orthopedic (Rehman, 2021 #171)
  * Pain scoring rate on numeric pain rating scale (NPRS) >3 during at least two activities (Rehman, 2021 #171)
  * Patients with positive Clarke's test/ Patellar grind test (Rehman, 2021 #171)
  * Pain while going up and down stairs, when sitting with knees flexed and with squatting, kneeling or returning from squat. (Powers, 2017 #172)

Exclusion Criteria:

* • Patients with other knee pathologies; meniscus tears, bursitis, patellar tendon injury, ligamentous injury

  * Degenerative joint disorders; knee osteoarthritis, rheumatoid arthritis etc.
  * Patellofemoral dislocation and / or frequent subluxation.
  * Patients having undergone lower extremity surgery
  * Those taking any pain medications

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
KOOS-PF Scale | 4 weeks
  KOOS-PF is a subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS) that specifically measures symptoms and function related to patellofemoral pain and osteoarthritis. It was developed to provide a more detailed assessment in this specific knee condition. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems. This direction, 100 indicating no problems.
Universal Goniometer | 4 weeks
  It has a scale for the measurement of the angle. The scale can extend from 0 to 180 degrees for half-circle models or 0 to 360 degrees for full-circle models.

CONTACTS AND LOCATIONS:
Overall Officials: Zunaira Saeed, Masters, Principal Investigator — University of Lahore; Umber Nawaz, PhD Scholar, Principal Investigator — University of Lahore; Ashfaq Ahmad, PhD, Study Chair — University of Lahore
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
After the completion of the study
Supporting Information: Study Protocol, SAP
Time Frame: After the completion of the study, tentatively in 2025
Access Criteria: by email